CLINICAL TRIAL: NCT06684353
Title: Clinical Presentation and Outcome of COPD Patients With Acute Exacerbation Attending Sohag University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mona Abdelaleem Hussien, Resident doctor at chest department Sohag University Hospital, Sohag University
Other Study IDs: Soh-Med-24-09-15MS
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients in ICU with high risk of mortality (non survivors): COPD patients on NIV / MV
- COPD patients in ICU with low risk of mortality ( survivors ): COPD patients on NIV / MV

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a worldwide public health challenge because of high prevalence and related disability and mortality (1).

Acute exacerbation of COPD (AECOPD), defned as the worsening of respiratory symptoms and requirement of additional clinical treatment, it reduces lung function and quality of life, and is accompanied by an increased disease-related burden, high hospital mortality and poor outcome (2).

Chronic obstructive pulmonary disease frequently coexists with other chronic diseases, namely comorbidities. They negatively impact prognosis, exacerbations and quality of life in COPD patients. Local and systemic inflammation have been proposed as having a potential role in explaining the association between COPD and these comorbidities (3).

ELIGIBILITY:
Inclusion Criteria:

patients with a confirmed COPD diagnosis according to (GOLD) guidelines, presented with acute exacerbation

Exclusion Criteria:

* Stable COPD
* Any other chronic chest diseases; Bronchial asthma or bronchiectasis

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients aged more than 18 years with a confirmed COPD diagnosis according to (GOLD) guidelines, presented with acute exacerbation
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-11-03 (Estimated); Study Completion 2025-11-03 (Estimated)

PRIMARY OUTCOMES:
Clinical Presentation and Outcome of COPD Patients With Acute Exacerbation Attending Sohag University Hospital | 1 year
  Detection which patient with COPD exacerbation has more risk of survival or mortality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fabbri LM, Boschetto P, Mapp CE; Global Initiative for Chronic Obstructive Lung Disease; Global Initiative for Asthma Management and Prevention. COPD guidelines: the important thing is not to stop questioning. Am J Respir Crit Care Med. 2007 Sep 15;176(6):527-8. doi: 10.1164/rccm.200706-854ED. No abstract available. PMID 17823358
- [Background] Bateman ED, Feldman C, O'Brien J, Plit M, Joubert JR; COPD Guideline Working Group of the South African Thoracic Society. Guideline for the management of chronic obstructive pulmonary disease (COPD): 2004 revision. S Afr Med J. 2004 Jul;94(7 Pt 2):559-75. PMID 15283307
- [Background] Corrections. Lancet Respir Med. 2017 Oct;5(10):e30. doi: 10.1016/S2213-2600(17)30336-3. Epub 2017 Sep 14. No abstract available. PMID 28918970
- [Background] Nakai T, Ueda M, Takeda R. Effects of calcium and magnesium ions on the interaction of corticosterone with rat brain cytosol receptor(s). Endocr Res Commun. 1978;5(2):81-90. doi: 10.3109/07435807809089010. PMID 102509
- [Background] Hand D. National Boards lose control of funding. Nurs Stand. 1991 Feb 13-19;5(21):20. No abstract available. PMID 1900164